CLINICAL TRIAL: NCT04736472
Title: Implementing Pharmacogenetic Testing in Gastrointestinal Cancers
Acronym: IMPACT-GI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Sony Tuteja, Principal Investigator, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UPCC 22220; 844763 (Other: University of Pennsylvania Perelman School of Medicine)
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Gastrointestinal Cancer
Keywords: Gastrointestinal Neoplasms; Fluorouracil; Capecitabine; Irinotecan; Fluoropyrimidines; Topoisomerase I inhibitors; Antimetabolites, Antineoplastics; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a nonrandomized, open-label study to investigate the feasibility of establishing and integrating a pharmacogenetic test into clinical oncology care. A historical control group of patients with gastrointestinal cancers enrolled in a biobank will be used to compare toxicity outcomes of the prospectively-genotyped patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- DPYD/UGT1A1 pharmacogenetic testing (Experimental): All patients will be screened for twelve single nucleotide polymorphisms (SNPs) in DPYD: DPYD*2A, *5, *6, *8, *9A, *10, *12, *13, rs2297595, rs115232898, rs67376798, HapB3.
  All patients will be screened for two SNPs in UGT1A1: UGT1A1*6, *28.
  Interventions: Device: Pharmacogenetic test

INTERVENTIONS:
Device: Pharmacogenetic test — Patients with reduced function alleles (DPYD intermediate or poor metabolizer and/or UGT1A1 poor metabolizer) will be recommended to receive dose reductions per clinical pharmacogenetic guidelines. Patients that do not carry actionable alleles (DPYD normal metabolizer and/or UGT1A1 normal or intermediate metabolizer) will receive standard dosing.

SUMMARY:
Pharmacogenomics (PGx) is the study of how genes affect a person's response to drugs. PGx testing for certain genes can help predict the risk of side effects from chemotherapy agents. Testing is not regularly performed in clinical practice due to long wait times for results and challenges with integrating test results in the electronic health record. Investigators leading this study hope to find out if providing cancer care providers with the ability to order a PGx test and electronically receive results with dosing recommendations will increase the use of these tests to guide treatment decisions and improve patient outcomes.

This is a non-randomized implementation study, which means that all participants in this study will undergo genotyping for a pharmacogenetic test. The investigators will primarily measure the feasibility of using this test to guide cancer care.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide informed consent
2. Male or female, aged 18 years or older at the time of study initiation
3. Pathologically confirmed gastrointestinal malignancy for which treatment with a fluoropyrimidine and/or irinotecan is indicated
4. Willing to undergo blood or saliva sampling for PGx testing and comply with all study-related procedures
5. Life expectancy of at least 6 months

Exclusion Criteria:

1. Prior treatment with irinotecan
2. DPYD or UGT1A1 genotype already known
3. Severe renal or hepatic impairment (or unacceptable laboratory values), including:

   * Neutrophil count of <1.5 x 109/L, platelet count of <100 x 109/L
   * Hepatic function as defined by serum bilirubin >1.5 x upper limit of normal (ULN), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) >2.5 x ULN, or in case of liver metastases ALT and AST>5 x ULN
   * Renal function as defined by serum creatinine >1.5 x ULN, or creatinine clearance <60 ml/min (by Cockcroft-Gault Equation)
4. Women who are pregnant or breast feeding, or subjects who refuse to use reliable contraceptive methods throughout the study
5. Treating physician does not want subject to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sony Tuteja, PharmD, MS, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol, SAP, ICF will be made available 1 year following enrollment of the last participant. IPD will be made available 6 months after publication of study results.
Access Criteria: Contact PI, Sony Tuteja, PharmD, sonyt@pennmedicine.upenn.edu with individual requests.

REFERENCES:
- [Derived] Varughese LA, Bhupathiraju M, Hoffecker G, Terek S, Harr M, Hakonarson H, Cambareri C, Marini J, Landgraf J, Chen J, Kanter G, Lau-Min KS, Massa RC, Damjanov N, Reddy NJ, Oyer RA, Teitelbaum UR, Tuteja S. Implementing Pharmacogenetic Testing in Gastrointestinal Cancers (IMPACT-GI): Study Protocol for a Pragmatic Implementation Trial for Establishing DPYD and UGT1A1 Screening to Guide Chemotherapy Dosing. Front Oncol. 2022 Jul 5;12:859846. doi: 10.3389/fonc.2022.859846. eCollection 2022. PMID 35865463

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 552 enrolled participants, 531 were eligible to begin study procedures.
Groups:
- Prospective Cohort: Enrollees were given DPYD and UGT1A1 testing before starting chemotherapy
- Confirmatory Cohort: Enrollees were given DPYD and UGT1A1 testing after starting chemotherapy at physician's request
- BioBank Control: Enrollees with biobank samples were tested for DPYD and UGT1A1 variants, and retrospectively chart reviewed for outcomes
Period: Overall Study
Arm/Group | Prospective Cohort | Confirmatory Cohort | BioBank Control
Started | 276 | 20 | 235
Completed PGx Testing | 268 | 20 | 231
Completed Relevant Chemotherapy | 225 | 20 | 229
Completed | 225 | 20 | 229
Not Completed | 51 | 0 | 6
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Protocol Violation | 48 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- BioBank Cohort: Enrollees with biobank samples were tested for DPYD and UGT1A1 variants, and retrospectively chart reviewed for outcomes
- Total: Total of all reporting groups
Arm/Group | Prospective Cohort | Confirmatory Cohort | BioBank Cohort | Total
Number analyzed (Participants) | 276 | 20 | 235 | 531
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 162 | 11 | 149 | 322
  >=65 years | 114 | 9 | 86 | 209
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 12 | 114 | 251
  Male | 151 | 8 | 121 | 280
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 0 | 1 | 10
  Not Hispanic or Latino | 265 | 19 | 0 | 284
  Unknown or Not Reported | 2 | 1 | 234 | 237
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 0 | 3 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 50 | 0 | 38 | 88
  White | 205 | 19 | 189 | 413
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 1 | 5 | 16
Region of Enrollment [Number; unit: participants]
  United States | 276 | 20 | 235 | 531
ECOG at Enrollment [Count of Participants; unit: Participants] — ECOG Performance Status from chart
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited self-care; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any self-care; totally confined to bed or chair
  5. Dead
  Participants
    0 | 151 | 12 | 102 | 265
    1 | 89 | 6 | 109 | 204
    2 | 20 | 1 | 21 | 42
    3 | 8 | 1 | 3 | 12
    NA | 8 | 0 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Number and Percentage of Participants Who Had Their Pharmacogenetic Tests Returned Prior to Initial Dose
Description: The Number and percentage of participants who had their pharmacogenetic tests returned prior to the first determined dose of chemotherapy.
Time Frame: 14 days
Population: Number and percentage of participants with both PGx test results and who began a qualifying chemotherapy. The BioBank Cohort and Confirmatory Cohort are not included in this measure as their PGx testing was intentionally ordered after their first dose of chemotherapy, therefore how many results were returned prior to first dose was not applicable.
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Cohort
Number analyzed (Participants) | 225
Participants
  PGx Result Returned before Chemotherapy | 130
  PGx Result Returned After Chemotherapy | 95

2. Primary Outcome: Fidelity: Level of Agreement With Dose Recommendations
Description: The number and percentage of participants with dose modifications made in agreement with the genotype-guided dosing recommendations for the first dose of chemotherapy.
Time Frame: 14 days
Population: Number and percentage of participants with an actionable genetic variant also receiving an interacting chemotherapy (DPYD Poor and Intermediate Metabolizers receiving fluoropyrimidine and UGT1A1 Poor Metabolizers receiving irinotecan). The BioBank Cohort and Confirmatory Cohort are not included in this measure as their PGx testing was intentionally ordered after their first dose of chemotherapy, therefore modifying their chemotherapy to match PGx results was not applicable.
Measure: Count of Participants; unit: Participants
Groups:
- Prospective Cohort: Enrollees were given PGx testing before starting 5-FU chemotherapy
Arm/Group | Prospective Cohort
Number analyzed (Participants) | 16
Participants
  Number and percent of participants with PGx test results returned before chemotherapy initiation | 11
  Number and percent of participants with DPYD dose mods in agreement to genotype-recommendations: number analyzed (Participants) | 6
  Number and percent of participants with DPYD dose mods in agreement to genotype-recommendations | 6
  Number and percent of participants with UGT1A1 dose mods in agreement to genotype-recommendations: number analyzed (Participants) | 5
  Number and percent of participants with UGT1A1 dose mods in agreement to genotype-recommendations | 5

3. Primary Outcome: Penetrance: Proportion of Pharmacogenetic Tests Ordered by Providers
Description: The number and percentage of participants with pharmacogenetic tests ordered compared to the number of patients eligible for testing at participating sites during the study timeframe
Time Frame: 14 days
Population: In order to calculate the penetrance of the intervention, as this was an implementation trial, it is necessary to consider the total number of patients who would have been eligible for recruitment. This includes both the prospective arms, as well as individuals in participating clinics during the study timeframe who were not approached for consent due to personnel and screening limitations.
Measure: Count of Participants; unit: Participants
Groups:
- Unique Patients Prescribed 5-FU: Total number of patients prescribed 5-FU chemotherapy at participating study sites during the timeframe number of individuals who would have been eligible for enrollment)
Arm/Group | Unique Patients Prescribed 5-FU
Number analyzed (Participants) | 1566
Participants | 288

4. Secondary Outcome: Severe Treatment Related Adverse Events (TRAE)
Description: Percentage of patients experiencing a severe TRAE (an event requiring hospitalization, emergency room visits, or oncology evaluation center). Severe TRAEs were one of the outcomes measured by the study.
Time Frame: 6 months
Population: Prospective and BioBank Cohorts are broken out into DGI and Non-DGI groups to compare participant outcomes by genotype.
Measure: Count of Participants; unit: Participants
Groups:
- Prospective Cohort, DGI Group: Enrollees were given DPYD and UGT1A1 testing before starting chemotherapy, and found to have a drug gene interaction (DGI) between their genotype and planned chemotherapy
- Prospective Cohort, Non-DGI Group: Enrollees were given DPYD and UGT1A1 testing before starting chemotherapy, and were not found to have a drug gene interaction (DGI) between their genotype and planned chemotherapy
- BioBank Cohort, DGI Group: Enrollees were tested for DPYD and UGT1A1 variants, and found to have a drug gene interaction (DGI) between their genotype and chemotherapy that would have been actionable, and retrospectively chart reviewed for outcomes
- BioBank Cohort, Normal Metabolizers Group: Enrollees were tested for DPYD and UGT1A1 variants, and were not found to have a drug gene interaction (DGI) between their genotype and chemotherapy, and retrospectively chart reviewed for outcomes
- Confirmatory Cohort: Enrollees were tested for DPYD and UGT1A1 variants after starting chemotherapy at physician request as a courtesy.
Arm/Group | Prospective Cohort, DGI Group | Prospective Cohort, Non-DGI Group | BioBank Cohort, DGI Group | BioBank Cohort, Normal Metabolizers Group | Confirmatory Cohort
Number analyzed (Participants) | 16 | 209 | 17 | 212 | 20
Participants
  Severe TRAEs | 6 | 63 | 10 | 66 | 10
  Treatment Modifications | 6 | 107 | 13 | 108 | 12
  Treatment Discontinuation | 5 | 49 | 8 | 60 | 8
Statistical Analysis 1: Comparison: Prospective Cohort, DGI Group vs BioBank Cohort, DGI Group; Severe TRAEs; Test type: Superiority; p = .224, Fisher Exact
Statistical Analysis 2: Comparison: BioBank Cohort, DGI Group vs BioBank Cohort, Normal Metabolizers Group; Severe TRAEs; Test type: Superiority; p = .025, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the first six cycles of chemotherapy, <6 months.
Description: Severe adverse events were defined as any related event requiring hospitalization, emergency room visits, oncology evaluation center care, or death. Other adverse events are all other adverse events that were collected that did not meet the serious criteria. Events were primarily assessed through medical records review.
Arm/Group | Prospective Cohort | Confirmatory Cohort | BioBank Cohort
All-Cause Mortality (participants affected / at risk) | 35/225 | 3/20 | 47/229
Serious Adverse Events (participants affected / at risk) | 69/225 | 10/20 | 76/229
Other Adverse Events (participants affected / at risk) | 214/225 | 20/20 | 140/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prospective Cohort (N=225) | Confirmatory Cohort (N=20) | BioBank Cohort (N=229)
Neutropenia (Blood and lymphatic system disorders) | 8 | 1 | 4
Diarrhea (Gastrointestinal disorders) | 13 | 4 | 16
Vomiting (Gastrointestinal disorders) | 15 | 2 | 19
Weakness (General disorders) | 10 | 0 | 0 — Not specifically assessed in the BioBank cohort, see other
Sepsis (Infections and infestations) | 7 | 1 | 11
Fever (General disorders) | 13 | 1 | 1
Thrombosis (Blood and lymphatic system disorders) | 10 | 0 | 0 — Not specifically assessed in the BioBank cohort, see other
Pain (General disorders) | 16 | 2 | 5
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 0 — Not specifically assessed in the BioBank cohort, see other
Other (General disorders) | 17 | 3 | 45
Nausea (Gastrointestinal disorders) | 14 | 2 | 16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prospective Cohort (N=225) | Confirmatory Cohort (N=20) | BioBank Cohort (N=229)
Neutropenia (Blood and lymphatic system disorders) | 98 | 13 | 47
Thrombocytopenia (Blood and lymphatic system disorders) | 91 | 8 | 22
Anemia (Blood and lymphatic system disorders) | 145 | 15 | 14
Diarrhea (Gastrointestinal disorders) | 115 | 11 | 40
Nausea (Gastrointestinal disorders) | 140 | 15 | 37
Vomiting (Gastrointestinal disorders) | 45 | 6 | 22
Mucositis (Gastrointestinal disorders) | 35 | 3 | 9
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 29 | 1 | 17
Heart Palpitations (Cardiac disorders) | 24 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 29 | 1 | 0
Peripheral Neuropathy (Nervous system disorders) | 0 | 0 | 33
Chest Pain (Cardiac disorders) | 14 | 1 | 5
Febrile Neutropenia (Blood and lymphatic system disorders) | 9 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/72/NCT04736472/Prot_SAP_001.pdf